CLINICAL TRIAL: NCT04092179
Title: Phase Ib/II Study of IDH2 Inhibitor Enasidenib in Combination With BCL2 Inhibitor Venetoclax in Patients With IDH2-Mutated Myeloid Malignancies (ENAVEN-AML)
Brief Title: Study of Enasidenib and Venetoclax in IDH2-Mutated Blood Cancers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Insufficient Funding
Sponsor: University Health Network, Toronto (Other)
Collaborators: Celgene (Industry); AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19-5939; ENAVEN-AML (Other: Princess Margaret Cancer Centre)
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Acute Myeloid Leukemia; Relapsed Cancer; Refractory Cancer; IDH2 Gene Mutation
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence; Neoplasms | interventions — enasidenib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venetoclax and Enadisenib (Experimental): Enasidenib and venetoclax will be taken by mouth (orally), once a day, every day, continuously.
  Every 28-day period will be called a cycle. Participants will start venetoclax alone on Cycle 1 Day 1 and continue the study drug alone until Day 15. On Day 15, participants will take enasidenib and venetoclax together and will continue to take the combination of study drugs until intolerable side effects or disease worsening.
  Interventions: Drug: Enasidenib; Drug: Venetoclax

INTERVENTIONS:
Drug: Enasidenib — Enasidenib is a drug that blocks a protein called isocitrate dehydrogenase (IDH) 2 from working. The family of IDH proteins have been indicated in the development of leukemia. By blocking IDH2, enasidenib may help stop cancer cells from growing. It is believed that the drug may be more useful in patients with a change (mutation) in their IDH 2 protein. The IDH2 gene (substances in the body that contain instructions for the proper development and function of cells) makes IDH2 proteins. As such, only patients with IDH 2 mutated gene are eligible for this study. Enasidenib is currently approved for the treatment of IDH2 mutated AML.
  Other Names: IDHIFA
Drug: Venetoclax — Venetoclax is a drug that blocks a protein called B-cell lymphoma (BCL2) protein from working. BCL2 is a protein that helps control whether a cell lives or dies and is thought to help cancer cells to live. Blocking BCL2 is believed to help kill cancer cells. Venetoclax is currently approved for the treatment of type of blood cancer called chronic lymphocytic leukemia (CLL) who have received prior treatment.
  Other Names: VENCLEXTA

SUMMARY:
The purpose of this research study is to see how safe and tolerable, and to find the highest or best dose, of an investigational combination of drugs called enasidenib and venetoclax, in patients with relapsed (the cancer has come back) or refractory (the cancer does not respond or have stopped responding to treatment) acute myeloid leukemia (AML, a type of blood cancer). This study will also see how useful the combination of enasidenib and venetoclax is in the treatment of patients with relapsed or refractory AML.

DETAILED DESCRIPTION:
This study will have two parts: Phase 1b and Phase 2. The part that patients may participate in will depend on when they join the study.

In the phase 1b portion of the study, small groups participants will receive increasing doses of venetoclax in combination with a flat dose of enadisenib until the highest dose or best dose of venetoclax that is safe and tolerable in combination with enadisenib is found.

In the phase 2 portion of the study, an additional group of participants will receive the highest or best dose of venetoclax found in the Phase 1b portion of the study with a flat dose of enadisenib to see how useful the combination is in treating relapsed or refractory acute myeloid leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance score of ≤2
* IDH2 (R140 or IDH R172) mutated AML disease status as determined by local laboratory
* Relapsed and/or refractory acute myeloid leukemia (AML). Treatment-naïve patients who are not eligible for standard induction chemotherapy or high-risk myelodysplastic syndromes (MDS) or myeloproliferative neoplasms (MPN) may also be eligible.
* Adequate hepatic function
* Adequate renal function
* Willing and able to provide informed consent
* In the absence of rapidly proliferative disease, the interval from prior treatment to time of initiation will be at least 7 days for cytotoxic and non-cytotoxic (immunotherapy) agents

Exclusion Criteria:

* Known allergy or hypersensitivity to enasidenib or venetoclax
* Previously received either an IDH2 inhibitor or BCL2 inhibitor
* With any uncontrolled clinically significant medical conditions
* The use of other chemotherapeutic agents or anti-leukemic agents, radiotherapy or other investigational therapy is not permitted during study with exceptions
* Receiving concomitant treatment with strong cytochrome P450 2A (CYP3A4) inhibitors within 3 days of start of study therapy
* Receiving concomitant strong CYP3A inducers (avasimibe, carbamazepine, phenytoin, rifampin, rifabutin, St. John's Wort) within 3 days of start of study therapy.
* Taking the following sensitive CYP substrate medications that have a narrow therapeutic range are excluded from the study unless the subject can be transferred to other medications at least 5 half-lives prior to the start of study treatment: paclitaxel and docetaxel (CYP2C8), phenytoin (CYP2C9), S-mephenytoin (CYP2C19), thioridazine (CYP2D6), theophylline, and tizanidine (CYP1A2)
* Active graft-versus-host-disease (GVHD) status post stem cell transplant
* Severe gastrointestinal or metabolic condition which could interfere with the absorption of oral study medications
* Concurrent active malignancy under treatment
* Administration or consumption of any of the following within 3 days prior to first dose of study drug: grapefruit or grapefruits products, Seville oranges (including marmalade containing Seville oranges) and start fruit
* Heart-rate corrected QT (QTc) interval ≥480 msec (Fridericia's formula) except for underlying right-bundle branch block (RBBB).
* Positive for HIV
* Subject has an unacceptable white blood cell count
* Positive urine pregnancy test,
* Participants who not willing to maintain adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 3 years
Dose Limiting Toxicity | 28 days
Maximum tolerated dose or Recommended Phase 2 Dose | 3 years
  Dose indicated by the mTPI decision
Duration of Response | 3 years
  The time from the date of first response until progression, relapse, death, or last follow-up.

SECONDARY OUTCOMES:
Overall Survival | 3 years
  The first day of treatment until death or last contact.
Event Free Survival | 3 years
  The number of days from the first day of treatment to the date of earliest evidence of relapse or progression, subsequent treatment other than stem cell transplant while in response, or death, or date of last disease assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Chan, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (2):
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Richard-Carpentier G, Gupta G, Koraksic C, Cathelin S, Wang L, Bankar A, Davidson M, Gupta V, Maze D, Minden MD, Murphy T, Schimmer AD, Schuh AC, Sibai H, Yee K, DiNardo CD, Brandwein J, McNamara CJ, Chan SM. Enasidenib plus venetoclax in patients with IDH2-mutated relapsed or refractory acute myeloid leukaemia or myelodysplastic syndrome (ENAVEN-AML): a multicentre, single-arm, phase 1b/2 trial. Lancet Haematol. 2025 Nov;12(11):e887-e897. doi: 10.1016/S2352-3026(25)00254-6. Epub 2025 Oct 8. PMID 41075807